CLINICAL TRIAL: NCT07312214
Title: A Randomized Controlled Trial of LED Red Light in Modulating Choroidal Microcirculation to Retard Retinal Atrophy in Pathological Myopia
Brief Title: LED Red Light in Modulating Choroidal Microcirculation to Retard Retinal Atrophy in Pathological Myopia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC-20250506-04
Record Dates: First submitted 2025-12-04; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Pathologic Myopia
Keywords: repeated low-level red light; LED; myopia; treatment
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): An RLRL device.
  Interventions: Device: LED red light
- Control (Sham Comparator): A sham RLRL device.
  Interventions: Device: Sham LED red light

INTERVENTIONS:
Device: LED red light — An RLRL device (660 nm, 65 mW/cm²). Twice daily, 3 minutes per session, 5 days per week, for a total duration of 12 months.
  Arms: Treatment
Device: Sham LED red light — A sham RLRL device (identical in appearance but delivering <10% of the original device's energy output) .
  Twice daily, 3 minutes per session, 5 days per week, for a total duration of 12 months.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if repeated low-level red light (RLRL) therapy works to treat pathologic myopia in adults. It will also learn about the safety of RLRL. The main questions it aims to answer are:

Does RLRL modulate choroidal microcirculation to retard retinal atrophy in pathological myopia? What medical problems do participants have when receiving RLRL therapy? Researchers will compare RLRL to a sham RLRL device (identical in appearance but delivering <10% of the original device's energy output) to see if RLRL works to treat pathologic myopia.

Participants will:

Take RLRL or sham RLRL twice daily, 3 minutes per session, 5 days per week, for a total duration of 12 months.

Visit the clinic once every 3 months for checkups and tests Keep a diary of their symptoms and their visual perception

DETAILED DESCRIPTION:
Pathological myopia (PM) is a major cause of irreversible visual impairment and blindness in adults, characterized by progressive axial elongation, choroidal thinning, impaired choroidal microcirculation, and subsequent retinal atrophy, which currently lacks effective therapeutic interventions. Against this clinical backdrop, this prospective randomized controlled trial is designed to systematically investigate the therapeutic efficacy and safety of repeated low-level red light (RLRL) therapy in adult patients with PM. The core research objectives are twofold: first, to verify whether RLRL can modulate choroidal microcirculatory function and thereby retard the progression of retinal atrophy in PM patients, and second, to comprehensively assess the safety profile of long-term RLRL administration by monitoring adverse events. To achieve these goals, the study will adopt a randomized controlled design, where eligible participants will be randomly assigned to either the active treatment group or the sham control group. The active treatment group will receive RLRL therapy, while the control group will be administered interventions using a sham RLRL device-this device is identical in appearance and operation mode to the active RLRL device but has an energy output of less than 10% of the original, aiming to exclude the placebo effect. The intervention regimen for both groups is standardized: participants will receive the assigned intervention twice daily, with each session lasting 3 minutes, 5 days per week, for a continuous 12-month course. During the study period, all participants will undergo regular follow-up visits at the clinic every 3 months, where a series of comprehensive assessments will be performed, including but not limited to visual acuity measurement, fundus examination, optical coherence tomography (OCT) for choroidal thickness and retinal structure evaluation, and choroidal blood flow dynamic detection to quantify microcirculatory changes. Additionally, participants will be instructed to maintain a detailed daily diary, recording the occurrence time, duration, and severity of any subjective symptoms (e.g., eye fatigue, photophobia) as well as changes in visual perception (e.g., contrast sensitivity, visual field changes), which will serve as supplementary data for safety monitoring and efficacy evaluation. Collectively, this study is expected to provide high-quality evidence for the clinical application of RLRL in the management of PM by clarifying its regulatory effect on choroidal microcirculation and its role in delaying retinal atrophy, while defining its safety boundaries.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18 to 55 years old;
* Baseline visual acuity: Best Corrected Visual Acuity (BCVA) ≥ 0.1 (LogMAR ≤ 1.0);
* Meeting the diagnostic criteria for high myopia: Spherical Equivalent (SE) ≤ -6.00 D and Axial Length (AL) ≥ 26.0 mm;
* Meeting one of the following pathological fundus changes:

  (i) Fundus manifestations corresponding to Category 2 (diffuse chorioretinal atrophy), Category 3 (patchy chorioretinal atrophy), or Category 4 (macular atrophy associated with choroidal neovascularization) of the META-PM classification criteria*; (ii) Category 1 of the META-PM classification criteria* complicated with macular schisis; (iii) BCVA < 0.6;

Exclusion Criteria:

* Concurrent with other ophthalmic diseases that may affect visual acuity or outcome assessment, including active myopic choroidal neovascularization (CNV) requiring anti-VEGF therapy, macular hole, vitreous hemorrhage, diabetic retinopathy, retinal detachment, retinal vein occlusion, optic neuritis, uveitis, severe cataract, and glaucoma;
* Systemic contraindications: Photosensitive epilepsy, autoimmune diseases (e.g., systemic lupus erythematosus), or pregnant/lactating women; Patients who have undergone intraocular surgery, laser treatment, or ophthalmic medication therapy within 3 months prior to enrollment;
* Patients unable to comply with regular follow-up (e.g., due to remote residence) or with cognitive impairment;
* Opaque refractive media that hinder fundus examination.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Choroidal vascular density | From enrollment to the end of treatment at 12 months
Choroidal vessel volume index | From enrollment to the end of treatment at 12 months

SECONDARY OUTCOMES:
Choroidal thickness | From enrollment to the end of treatment at 12 months
Distance between Bruch's membrane and choroidal-scleral interface | From enrollment to the end of treatment at 12 months
Retinal thickness | From enrollment to the end of treatment at 12 months
Retinal vascular density | From enrollment to the end of treatment at 12 months
Proportion of participants developed diffuse chorioretinal atrophy | From enrollment to the end of treatment at 12 months

OTHER OUTCOMES:
Changes in BCVA | From enrollment to the end of treatment at 12 months
  best-corrected visual acuity
Incidence of allergic reactions | From enrollment to the end of treatment at 12 months
  including photophobia, blurred near vision, afterimage, elevated IOP, headache, nausea, and vomiting
Changes in AL | From enrollment to 12-month
  axial length
Changes in SE | From enrollment to the end of treatment at 12 months
  spherical equivalent
Changes in IOP | From enrollment to the end in 12-month
  intra ocular pressure
Changes in VF | From enrollment to the end of treatment in 12-month
  visual field, using microperimetry

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Disease Prevention and Treatment Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
After the completion of the study, all individual participant data (IPD), including clinical examination data, demographic information, and other relevant datasets, will be shared upon legitimate and reasonable requests following rigorous anonymization procedures to protect participant privacy.